CLINICAL TRIAL: NCT05210309
Title: National Project to Implement Mesenchymal Stem Cell for the Treatment of Perianal Crohn's Fistula (the PRIME Study)
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Hospital Universitario Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Jose-M Ramirez, Profesor, Universidad de Zaragoza
Other Study IDs: UZaragoza-1
Record Dates: First submitted 2021-12-29; First posted 2022-01-27 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Safety; Efficacy, Self

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Stem Cell Therapy — Application of Darvadstrocel locally, after fistula tract curettage and internal opening closure.
  Other Names: Darvadstrocel

SUMMARY:
Darvadstrocel is an expanded allogeneic adipose-derived mesenchymal stem cell therapy for the treatment of complex perianal fistulas in patients with Crohn's disease. Safety and efficacy of the procedure has been sufficiently demonstrated and the Spanish Agency of Medication approved its application a few months ago. Being aware about the difficulties to a proper application and management of the stem cells the Spanish Stem Cell therapy group devised, in a joint activity with the Spanish Group GERM (Grupo Español de Rehabilitacion Multimodal) dedicated to expand the best surgical clinical practices, a national project for the application of the therapy. The objective is to get a homogeneous implementation in all hospitals in Spain that have being baked to use this biological therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older who have complex perianal Crohn ﬁstula
* non-active or mildly active luminal Crohn's disease for at least 6 months.
* The ﬁstula had to have been draining for at least 6 weeks before inclusion.

Exclusion Criteria:

• Patient with recto-vaginal ﬁstula; rectal or anal stenosis; or active severe proctitis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patiens with perianal Crohn´s Disease who do not respond to current therapies.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Therapeutic Efficacy of Darvadstrocel-Clinical | 6 moths
  Clinical closure of the Fistula
Therapeutic Efficacy of Darvadstrocel-MRI | 6 moths
  MRI imaging closure of the Fistula

SECONDARY OUTCOMES:
Quality of Life (QoL) | 6 moths
  QoL according to dedicated questionnaire (EuroQoL 5D-3L)
PATIENT REPORTED OUTCOMES (PROs) | 6 moths
  A Dedicated self complementary questionnaire (PROMs)
Efficiency | 6 moths
  Cost-Effectiveness of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jose-M Ramirez, Prof, Principal Investigator — Catedra GERM Medicina Perioperatoria; Damian Garcia-Olmo, Prof, Study Chair — Fundación Jiménez Diaz. Madrid
Locations (4):
- Spain (4):
  - Hospital de Elche, Elche, Alicante
  - HOSPITAL Meixoeiro Vigo, Vigo, Pontevedra
  - Hospital Vall D´Hebron, Barcelona
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott LJ. Darvadstrocel: A Review in Treatment-Refractory Complex Perianal Fistulas in Crohn's Disease. BioDrugs. 2018 Dec;32(6):627-634. doi: 10.1007/s40259-018-0311-4. PMID 30298387
- [Background] Panes J, Rimola J. Perianal fistulizing Crohn's disease: pathogenesis, diagnosis and therapy. Nat Rev Gastroenterol Hepatol. 2017 Nov;14(11):652-664. doi: 10.1038/nrgastro.2017.104. Epub 2017 Aug 9. PMID 28790453
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Diez MC, Tagarro I, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Long-term Efficacy and Safety of Stem Cell Therapy (Cx601) for Complex Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2018 Apr;154(5):1334-1342.e4. doi: 10.1053/j.gastro.2017.12.020. Epub 2017 Dec 24. PMID 29277560
- [Result] Garcia-Olmo D, Gilaberte I, Binek M, D Hoore AJL, Lindner D, Selvaggi F, Spinelli A, Panes J. Follow-up Study to Evaluate the Long-term Safety and Efficacy of Darvadstrocel (Mesenchymal Stem Cell Treatment) in Patients With Perianal Fistulizing Crohn's Disease: ADMIRE-CD Phase 3 Randomized Controlled Trial. Dis Colon Rectum. 2022 May 1;65(5):713-720. doi: 10.1097/DCR.0000000000002325. PMID 34890373
- [Result] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896